CLINICAL TRIAL: NCT04971629
Title: A Prospective Observational Study of the Relationship Between Cannabis Use, Biomarkers, Tissue Cannabinoid Levels and Clinical Outcomes in Patients With Osteoarthritis
Brief Title: The Relationship Between Cannabis Use, Biomarkers, Tissue Cannabinoid Levels and Clinical Outcomes in Patients With OA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Hance Clarke, Director Pain Services, Toronto General Hospital, University Health Network, Toronto
Other Study IDs: 20-5918 OA
Record Dates: First submitted 2021-06-29; First posted 2021-07-21 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Osteo Arthritis Knee

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Patients with knee osteoarthritis who use medical cannabis to manage MSK symptoms.
- Cohort 2: Patients with knee osteoarthritis who do not use medical cannabis.

SUMMARY:
Osteoarthritis (OA), the most common form of arthritis, is a leading cause of disability, affecting the quality of life, pain, and physical functioning of 4.6 million Canadians. About half of OA patients have limited response to primary therapy. The number of OA patients continues to rise, affecting the quality of life of those with OA. There is a dire need to develop future effective treatment options. Cannabis is a potential therapy for those with OA and may provide analgesic, anti-inflammatory, and disease modifying effects. The common barriers to use are a lack of knowledge regarding efficacy, access, and commonly used products, doses and routes of administration. No high-quality clinical trials of cannabis for OA have been conducted, leaving physicians struggling to guide and inform patients regarding symptom relief. Findings from clinical trials of cannabis for other painful conditions have been variable, perhaps due to suboptimal cannabis products and failure to consider important patient characteristics. The goal of the current study is to characterize patient- and cannabis-level factors that are associated with OA pain and address other knowledge gaps.

DETAILED DESCRIPTION:
Given the heterogeneity of OA, it is likely that any therapeutic (or harmful) effect of cannabis will vary based on patient characteristics and levels of cannabinoids in the cannabis product used. In this study, the investigators will measure the association between patient- and cannabis-level characteristics and patient outcomes among OA patients who use cannabis to manage their MSK symptoms and those who do not. 1) A number of patient-level factors are capable of modulating the symptoms and pathology of OA. These include microRNAs (miRNAs), metabolites, and cytokines/growth factors. Alterations in these molecules have been detected in the blood of patients with OA and thus are potential biomarker candidates of disease, prognosis or even therapeutic efficacy. Biomarkers will be measured in a cohort of patients with OA to investigate whether they predict the perceived effectiveness of cannabis and whether they differ among cannabis users and non-users. In addition, the investigators will look at the correlation between biomarker(s) levels and patients' reported outcomes among cannabis users vs non-users. 2) Chondrocytes from OA joints express a wide range of cannabinoid receptors, so there is the promise that these cells could respond to cannabinoid-based medicines. In a subset of cannabis users, tissue samples from the knee will be collected to determine if the products being consumed penetrate the tissues. 3) Due to the varied chemical constituents in cannabis products, and the lack of clear understanding of the pharmacological effects of hundreds of varieties of medical cannabis, there is a need for in-depth investigations into cannabis strains produced in Canada and those consumed by patients. Research led by our group found that industry products vary from batch to batch and labeling can be inaccurate, highlighting the need for further investigation into the relationship between cannabis' chemical constituents and its clinical effect.

A total of 1200 adults with knee osteoarthritis, 600 participants who use medical cannabis to manage their symptoms and 600 who do not use it will be included. All participants will complete a set of questionnaires that will collect information about demographics, medical condition(s), current pharmaceutical pain management, and cannabis use (if any). In addition, these questionnaires will evaluate pain severity and the impact of pain on day-to-day life, anxiety, depression, and quality of life. Participants will also be required to provide a blood sample to identify biomarkers. An additional blood sample will be collected from participants who use cannabis to measure level of cannabinoids in the blood. In a subset of 105 participants (100 cannabis users and 5 cannabis non-users) undergoing total knee replacement surgery, samples of tissue discarded during surgery will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥25
2. Able to understand and read English
3. Diagnosed with knee OA or seeking treatment for knee related OA
4. Experienced pain in the knee on most days for at least 3 months

Exclusion Criteria:

1. Used cannabis recreationally, but not medically in the past 3 months.
2. Total joint arthroplasty (TJA) within a year of informed consent.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with knee osteoarthritis (n=600 cannabis users and n=600 cannabis non-users); a subset of the cannabis users (n=100) and cannabis non-users (n=5) will be undergoing total knee replacement surgery.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2021-07-13 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
MicroRNAs (Using Next Generation Sequencing) | Baseline
  Next Generation Sequencing will be used to identify differentially expressed circulating miRNAs in plasma samples.
Cytokines (High-throughput Luminex-based assays) | Baseline
  High-throughput ELISA methodology will be used to determine levels of circulating inflammatory cytokines. Cytokines of interest include interferon (IFN)y, interleukin (IL)-1ß, IL-6, IL-8, IL-10, macrophage inflammatory protein (MIP)-1b, tumor necrosis factor (TNF)α], and metabolic cytokines (Leptin and adiponectin).
Pain Mediators (High-throughput Luminex-based assays) | Baseline
  High-throughput ELISA methodology will be used to determine levels of circulating pain mediators. Pain mediators of interest include prostaglandin(PG)E2 and nerve growth factor (NGF).
Metabolites (Metabolomics Analyses) | Day of Surgery
  A high throughput metabolomics approach will be used to determine differences in the circulating metabolites that may contribute to patient response to cannabis.

SECONDARY OUTCOMES:
Pain Disability Index (PDI) | Baseline
  The PDI measures the degree to which aspects of a patient's life are disrupted by chronic pain. Patients indicate the overall impact of pain on 7 categories in their life (family/home responsibilities; recreation; social activity; occupation; sexual behaviour; self-care; life-support activities) on a scale from 0 (no disability) to 7 (worst disability). The PDI has good reliability and validity, with moderate test-retest reliability.
Patient Health Questionnaire (PHQ-8) | Baseline
  The PHQ-8 is a self-administered version of the PRIME-MD diagnostic instrument for common mental disorders. The PHQ-8 is an adaptation of PHQ-9 depression module which scores the DSM-IV criteria as "0" (not at all) to "3" (nearly every day). The item9 "How often during the past 2 weeks were you bothered by thoughts that you would be better off dead, or of hurting yourself in some way?", was deleted. The eight-item PHQ is established as a valid diagnostic and severity measure for depressive disorders in large clinical studies.
Generalized Anxiety Disorder Assessment (GAD-7) | Baseline
  The GAD-7 is a measure of anxiety symptoms and a screening tool for generalized anxiety disorder (GAD). This 7-item scale assesses signs of GAD (e.g. "Feeling afraid as if something awful might happen") with response options of: (1) Not at all, (2) Several days, (3) More than half the days, (4) Nearly every day. The GAD-7 is frequently used in primary and outpatient care populations and has been found to have adequate validity and good reliability.
Patient-Reported Outcomes Measurement Information System (PROMIS) - Pain Interference - Short Form 8a | Baseline
  This instrument assesses the self-reported impact of pain on daily activities, social, emotional, physical, and recreational activities. This measure assesses pain interference over the past 7 days. Each of 8 items is rated on a scale of 1-5 (1=not at all, 2=a little bit, 3=somewhat, 4=quite a bit, and 5=very much).
Numeric Rating Scale (NRS)- Pain Intensity/Severity | Baseline
  This is a custom designed questionnaire containing 4 questions to assess the intensity/severity of the pain. The11-point NRS (0-10) with end points labeled "0=no pain" and "10=pain as bad as you can imagine" to measure the intensity/severity of the "worst", "least", "average" and "now" (present) pain.
Quality of Life Scale (QoLS) | Baseline
  This is a custom designed questionnaire with only one item developed based on the final question of EuroQol-5D-5L to rate how "good or bad your health is TODAY" by selecting one number on the line corresponding to his/her perceived health. This 11point numeric rating scale with the endpoints labeled "0= Worst imaginable health state" and "10= Best imaginable health state."
Ultra-performance liquid chromatography/mass spectrometry (UPLC/MS) | Day of Surgery
  The chemical composition of the cannabis samples provided by participants will be analyzed using UPLC/MS. This instrumentation will also be used to identify the level of phytocannabinoids within the blood of each cannabis user and, in a subset of 100 patients, undergoing total knee arthroplasty, joint tissue will be analyzed for the presence/absence of phytocannabinoids as well.

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No